CLINICAL TRIAL: NCT02435992
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Oral RPC1063 as Induction and Maintenance Therapy for Moderate to Severe Ulcerative Colitis
Brief Title: Safety and Efficacy Trial of RPC1063 for Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPC01-3101
Record Dates: First submitted 2015-04-24; First posted 2015-05-06 (Estimated); Results first posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ozanimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RPC1063 (Ozanimod) (Experimental): 1mg, daily oral administration during Induction and Maintenance periods.
  Interventions: Drug: RPC1063
- Placebo (Placebo Comparator): Daily oral administration during Induction and Maintenance periods.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RPC1063
  Arms: RPC1063 (Ozanimod)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether RPC1063 is effective in the treatment of Ulcerative Colitis (UC).

DETAILED DESCRIPTION:
The trial is composed of 2 periods: Induction and Maintenance. In the Induction Period (IP), patients will be entered into the trial in 2 separate cohorts (Cohort 1 and Cohort 2).Patients from Cohort 1 and 2 in clinical response at the end of the IP will proceed through to the Maintenance Period (MP). Patients from Cohort 1 and 2 who participate in this trial may also qualify to participate in an optional Open-Label Extension (OLE) trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years (at screening for Cohort 1 and 2)
* UC confirmed on endoscopy
* Moderately to severely active UC (May score 6-12)
* Currently receiving treatment with aminosalisylate, prednisone, or budesonide
* Can be receiving azathioprine, mercaptopurine, or methotrexate, but treatment will be stopped prior to randomization

Exclusion Criteria:

* Have severe extensive colitis as evidence by:
* Physician judgment that the patient is likely to require colectomy or ileostomy within 12 weeks of baseline.
* Current or recent (within 3 months) evidence of fulminant colitis, toxic megacolon, or bowel perforation.
* Diagnosis of CD, indeterminate colitis, or the presence of fistula consistent with CD or microscopic colitis, radiation colitis, or ischemic colitis
* Clinically relevant cardiovascular conditions or other relevant diseases that could impact the implementation or interpretation of the trial, or put the patient at risk
* History of uveitis or unknown macular edema
* Pregnancy, lactation, or a positive serum β-human chorionic gonadotropin (β-hCG) measured during screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2015-06-17 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AnnKatrin Petersen, M.D., MSc., Study Director — Celgene
Locations (372):
- United States (113):
  - Arizona Digestive Health, Sun City, Arizona
  - Adobe Clinical Research LLC, Tucson, Arizona
  - Arkansas Gastroenterology, P.A., North Little Rock, Arkansas
  - Anaheim Clinical Trials, Anaheim, California
  - Aurora Care Clinic, Costa Mesa, California
  - Valley View Internal Medicine, Garden Grove, California
  - Davita Clinical Trials, LLC, Huntington Beach, California
  - University of California San Diego Medical Center, La Jolla, California
  - OM Research, Lancaster, California
  - University of Southern California - Keck School of Medicine, Los Angeles, California
  - Southern California Research Institute Medical Group, Inc., Los Angeles, California
  - Gastrointestinal Biosciences, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Facey Medical Foundation (Parent), Mission Hills, California
  - Alliance Clinical Research, LLC, Oceanside, California
  - Medical Associates Research Group, Inc., San Diego, California
  - University of California at San Francisco (PARENT), San Francisco, California
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Gastro Florida, Clearwater, Florida
  - Clinical Research of West Florida Inc - Clearwater, Clearwater, Florida
  - Advanced Pharma Research, Inc, Delray Beach, Florida
  - Universal Axon Clinical Research, Doral, Florida
  - Dolphin Medical Research, Doral, Florida
  - South Florida Clinical Trials, Hialeah, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - City Medical Group, Miami, Florida
  - Advanced Clincial Research, Miami, Florida
  - Advanced Clinical Research of Miami, Miami, Florida
  - Regenerate Clinical Trials, Miami, Florida
  - Advanced Research for Health Improvement, Naples, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - NSB Research, New Smyrna Beach, Florida
  - Harmony Clinical Research, North Miami Beach, Florida
  - Med-Care Research, North Miami Beach, Florida
  - Center For Digestive Health, Orlando, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - DBC Research, Corp, Pembroke Pines, Florida
  - Theia Clinical Research, LLC, Pinellas Park, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Atlanta Gastroenterology Associates LLC, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - Northwestern University Feinberg Sch of Medicine Division of Gastroenterology, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - DM Clinical Research, Oak Lawn, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - University of Maryland Medical Group, Baltimore, Maryland
  - Woodholme Gastroenterology, Baltimore, Maryland
  - Johns Hopkins Clinical Research Network, Baltimore, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Charm City Research Group, Towson, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Commonwealth Clinical Studies, PLLC., Brockton, Massachusetts
  - Community Clinical Research Network, Marlborough, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Center For Digestive Health, Troy, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Ehrhardt Clinical Research, LLC, Belton, Missouri
  - Clinical Research Professionals, LLC - De Paul Medical Dr, Bridgeton, Missouri
  - Mercy Research, Springfield, Missouri
  - Washington University, St Louis, Missouri
  - Clinical Research Professionals LLC - The Pines Court, St Louis, Missouri
  - Clinical Research Professionals, LLC - Olde Cabin Rd, St Louis, Missouri
  - Mary Hitchcock Memorial Hospital, Lebanon, New Hampshire
  - NY Scientific, Brooklyn, New York
  - Long Island Clinical Research Associates, Great Neck, New York
  - Icahn School of Medicine Mount Sinai Beth Isreal, New York, New York
  - Concord Medical Group PRIME, New York, New York
  - New York University School of Medicine, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai - PRIME, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas HealthCare System Digestive Health, Charlotte, North Carolina
  - East Carolina Gastroenterology, PA, Jacksonville, North Carolina
  - Kinston Medical Specialists, PA, Kinston, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - UC Health Clinical Trials Office, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Clinical Trials Management Office, Columbus, Ohio
  - Clinical Inquest Center Ltd, Springfield, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Digestive Disease Specialists, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Consultants in Gastroenterology, PA, Columbia, South Carolina
  - Gastroenterology Associates of Orangeburg, Orangeburg, South Carolina
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - Brooke-Army Medical Center, Fort Sam Houston, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Gulf Coast Research Group LLC, Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - Houston Endoscopy and Research Center, Houston, Texas
  - Gastroenterology Research of San Antonio, LLC, San Antonio, Texas
  - San Antonio Gastroenterology, San Antonio, Texas
  - Texas Digestive Disease Consultants - Southlake, Southlake, Texas
  - Spring Gastroenterology, Spring, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Gastroenterology, LTD, Virginia Beach, Virginia
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Argentina (5):
  - Hospital Italiano, Buenos Aires
  - Instituto DAMIC Fundacion Rusculleda, Córdoba
  - Hospital Italiano de La Plata, La Plata
  - Instituto Medico CER, Quilmes
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario
- Australia (9):
  - Centre For Digestive Diseases, Five Dock, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Cabrini Hospital Malvern, Malvern, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Monash Medical Centre Clayton, Bentleigh East
  - Royal Prince Alfred Hospital, Camperdown
- Medical University Vienna, Vienna, Austria
- Belarus (3):
  - Gomel Regional Clinical Hospital, Homyel
  - City Clinical Hospital No 10, Minsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
- Belgium (5):
  - Imeldaziekenhuis, Bonheiden
  - AZ Maria Middelares, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - CHC - Clinique St-Jospeh, Liège
- Bulgaria (15):
  - Medical Centre "Asklepii", OOD, Dupnitsa
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - UMHAT "Kaspela", EOOD, Plovdiv
  - MC Rusemed ltd., Rousse
  - NMTH "Tsar Boris III", Sofia
  - MHAT "Lyulin", EAD, Sofia
  - City Clinic UMHAC EOOD, Sofia
  - MHAT 'Tokuda Hospital Sofia', EAD, Sofia
  - UMHAT 'Tsaritsa Yoanna - ISUL', EAD, Sofia
  - Fourth MHAT - Sofia EAD, Sofia
  - UMHAT 'Sveta Anna' AD, Sofia
  - UMHAT "SofiaMed", OOD, Sofia
  - Medical Center "Nov Rehabilitatsionen Tsentar", EOOD, Stara Zagora
  - MHAT 'Sv. Marina', EAD, Varna
  - MC Medica Plus, Veliko Tarnovo
- Canada (12):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Brandon Medical Arts Clinic, Brandon, Manitoba
  - Viable Clinical Research - Lindsay, Lindsay, Ontario
  - LHSC - University Hospital, London, Ontario
  - LHSC - Victoria Hospital, London, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Toronto Digestive Disease Associates, Inc., Vaughan, Ontario
  - Centre integre de sante et de services sociaux de la Monteregie-Centre - Hopital Charles-Le Moyne, Greenfield Park, Quebec
  - The Ottawa Hospital - General Campus, Ottawa, Quebec
  - CHUS - Hôpital Fleurimont, Sherbrooke, Quebec
- Croatia (5):
  - Clinical Hospital Center Osijek, Osijek
  - Clinical Hospital Centre Rijeka, Rijeka
  - Clinical Hospital "Sveti Duh", Clinic of Internal Diseases, Zagreb
  - Clinical Hospital Center Sestre milosrdnice Clinic of Internal Diseases, Zagreb
  - Clinical Hospital Dubrava, Clinic of Internal Medicine, Department of Gastroenterology, Zagreb
- Czechia (9):
  - Vojenska nemocnice Brno, Brno
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - GASTRO JeKa s.r.o., Klatovy
  - Gregar s.r.o., Olomouc
  - PreventaMed, Olomouc
  - Institut klinicke a experimentalni mediciny, Prague
  - Thomayerova nemocnice, Prague
  - ISCARE, a.s., Prague
  - Nemocnice Slany, Slaný
- Georgia (5):
  - LTD Research Institute of Clinical Medicine, Tbilisi
  - LLC Vivamedi, Tbilisi
  - LTD Academician N.Kipshidze Central University Clinic, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - LTD Coloproctological Center, Tbilisi
- Germany (16):
  - Charite - Universitaetsmedizin Berlin Charité - Campus Benjamin Franklin, Berlin
  - Charite - Campus Virchow-Klinikum, Berlin
  - DRK Kliniken Berlin Westend, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Medical Care Unit Dachau, Dachau
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Crohn Colitis Centrum Rhein Main, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - EUGASTRO GmbH, Leipzig
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Universitatsklinikum Ulm, Ulm
- Greece (5):
  - Laiko General Hospital of Athens, Athens
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Larissa, Larissa Thessaly
  - General Hospital of Thessaloniki Hippokration, Thessaloniki
  - 424th Army General Hospital, Thessaloniki
- Hungary (14):
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - Bekes Megyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaz, Békéscsaba
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Semmelweis Egyetem, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Szent Margit Korhaz, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza, Gyula
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Vasutegeszsegugyi Kft. - Debreceni Egeszsegugyi Kozpont, Létavértes
  - Mohacsi Korhaz, Mohács
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Israel (6):
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (12):
  - Azienda Ospedaliera Universitaria Policlinico Sant Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli Presidio Ospedale Sacco, Milan
  - A.O.U. Policlinico di Modena, Modena
  - Azienda Socio Sanitaria Territoriale di Monza (Presidio San Gerardo), Monza
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Complesso Integrato Columbus, Roma
  - Istituto Clinico Humanitas, Rozzano (MI)
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo FG
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Moldova (4):
  - "Sfanta Treime" Clinical Municipal Hospital, Chisinau
  - Clinical Hospital of the Ministry of Health, Department of Endoscopic Surgery, Chisinau
  - "Sf. Arhanghel Mihail" Municipal Clinical Hospital, Chisinau
  - Republican Clinical Hospital, Chisinau
- Netherlands (6):
  - Vrije Universiteit Medisch Centrum (VUMC), Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen (UMCG), Groningen
  - Maastricht University Medical Center, Maastrich
  - Zuyderland Medisch Centrum - Sittard-Geleen, Sittard-Geleen
  - ETZ Elisabeth, Tilburg
- New Zealand (2):
  - Christchurch Hospital NZ, Christchurch
  - Dunedin Public Hospital, Dunedin
- Poland (17):
  - Clinsante S.C. Osrodek Badan Klinicznych, Bydgoszcz
  - Specjalistyczna Przychodnia Lekarska Medicus, Chorzów
  - PLEJADY Sp. z o.o. (LLC) Medical Centre, Krakow
  - Centrum Medyczne A-Z Clinic, Krakow
  - Healthcare Center Orkan Med Stec Michalska Spolka Jawna, Ksawerów
  - GLOBE Clinical Research Sp. z o.o. LLC, Kłodzko
  - Santa Familia Centrum Badan, Profilaktyki i Leczenia, Lodz
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - Trialmed Llc, Piotrkow Trybunalski
  - SOLUMED Centrum Medyczne, Poznan
  - Specjalistyczna Praktyka Lekarska dr med. Marek Horynski, Sopot
  - KO-MED Centra Kliniczne Staszow, Staszów
  - GASTROMED Kopon, Zmudzinski and Partners Specialist Centre for Gastroenterology and Endoscopy, Spe, Torun
  - MDM Healthcare Centre, Warsaw
  - Nzoz Vivamed, Warsaw
  - Health Centre Metabolic Diseases Outpatient Clinic in Wierzchoslawice, Wierzchosławice
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
- Romania (7):
  - Bacau County Emergency Hospital, Department of Gastroenterology, Bacau
  - Hyperclinica MedLife Grivita, Bucharest
  - Bucharest University Emergency Hospital, Department of Internal Medicine II, Bucharest
  - TVM MED SERV SRL, Medical Center for Gastroenterology, Hepatology and Digestive Endoscopy, Cluj-Napoca
  - Sf. Apostol Andrei Constanta Emergency Clinical County Hospital, Constanța
  - Craiova County Emergency Clinical Hospital, Craiova
  - "Pius Brinzeu" County Emergency Clinical Hospital, Department of Gastroenterology and Hepatology, Timișoara
- Russia (20):
  - Multidisciplinary Medical Clinic "Anthurium", Barnaul
  - Road Clinical Hospital on Station Irkutsk-Passazhirskiy of OJSC Russian Railways, Irkutsk
  - SBEI HPE "Kazan State Medical University" of the MoH of the RF, Kazan'
  - FSBIH "Central Clinical Hospital of Russian Academy of Sciences", Moscow
  - SBIH of Nizhniy Novgorod region " Nizhniy Novgorod Regional Clinical Hospital n.a. N.A. Semashko", Nizhny Novgorod
  - SBEIHPE Novosibirsk State Medical University, Novosibirsk
  - FSBI "Scientific Research Institute of Physyology and Basic Medicine" under the SB of RAMS, Novosibirsk
  - BHI of Omsk region "Clinical Oncology Dispensary", Omsk
  - SBEI HPE Rostov State Medical University of the MoH of the RF, Rostov-on-Don
  - SPb SBIH Alexandrovskaya City Hospital, Saint Petersburg
  - FFSBI "The Nikiforov Russian Center of Emergency and Radiation Medicine", Saint Petersburg
  - FSMEI HPE "Military Medical Academy n.a. S.M.Kirov"of Ministry of Defense of Russia, Saint Petersburg
  - SBIH City Clinical Hospital #31, Saint Petersburg
  - SPb SBIH City Hospital # 26, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Union Clinic, Saint-Peterburg
  - Private Educational Institution of Higher Education "Medical University "REAVIZ", Samara
  - LLC Medical Company Hepatologist, Samara
  - SBEI HPE "Stavropol State Medical Academy" MoH of RF, Stavropol
  - Regional Clinical Hospital, Vladimir
- Serbia (8):
  - Clinical Hospital Center Bezanijska Kosa, Clinic of Internal Medicine, Belgrade
  - Clinical Center of Serbia, Clinic of Gastroenterology and Hepatology, Department of Gastroenterology, Belgrade
  - Clinical Hospital Center Zvezdara Clinic of Internal Diseases, Belgrade
  - Military Medical Academy, Clinic of Gastroenterology and Hepatology, Belgrade
  - Clinical Hospital Center Zemun Department of Gastroenterology, Belgrade
  - Clinical Center Kragujevac, Clinic of Internal Medicine, Center for Gastroenterohepatology, Kragujevac
  - Clinical Center Nis, Clinic of Gastroenterology and Hepatology, Niš
  - General Hospital Djordje Jovanovic Zrenjanin, Zrenjanin
- Slovakia (11):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta, Banská Bystrica
  - Alian s.r.o., Bardejov
  - PRO SANUS, a.s., Poliklinika ProCare Central, Bratislava
  - IBDcentrum s.r.o., Bratislava
  - Slovak Research Center-team member, Sukromna gastroenterologicka ambulancia, Ilava
  - Gastroped s.r.o., Košice
  - Gastroeneterologicka ambulancia MUDr. Peter Hegyi, s.r.o., Malacky
  - PIGEAS s.r.o., Martin
  - Nemocnica s poliklinikou S. Kukuru Michalovce, a.s., Michalovce
  - Gastromedic s.r.o., Nové Zámky
  - EndoCorp s.r.o., Trnava
- South Africa (6):
  - Dr MJ Prins Practice, Cape Town
  - Tiervlei Trial Centre, Cape Town
  - Endocare Research, Cape Town
  - Dr JP Wright Practice, Cape Town
  - Dr YS Nanabhay Practice, Johannesburg
  - Emmed Research, Pretoria
- South Korea (16):
  - Inje University Haeundae Paik Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Konyang University Hospital, Daejeon
  - Hanyang Univerisy Guri Hospital, Guri-si
  - Seoul National University Bundang Hospital, Seongnam
  - CHA Bundang Medical Center CHA University, Seongnam-si
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - The Catholic University of Korea, St.Vicent's Hospital, Suwon
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (4):
  - University Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - University Hospital of the Canary Islands (HUC) La Laguna, San Cristóbal de La Laguna
  - University Hospital Virgen del Rocio, Seville
- Ukraine (29):
  - RCI Chernivtsi Regional Clinical Hospital Dept of Gastroenterology Bukovinsky SMU, Chernivtsi
  - Dnipropetrovsk I.I. Mechnykov Regional Clinical Hospital, Dnipropetrovsk
  - Si Institute Of Gastroenterology Of Namsu Dept Of Stomach And Duodenum Diseases, Dnipropetrovsk
  - Ivano-Frankivsk City Clinical Hospital #1 Dep of Surgery SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - Central City Clinical Hospital Dept of Theraphy No. 2 SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - CI of PH Kharkiv CCH #2, Kharkiv
  - GI L.T.Malaya Therapy National Institute of the NAMS of Ukraine, Kharkiv
  - Kyiv City Clinical Hospital #1, Kyiv
  - SI Republican Clinical Hospital of the MOHU Dept of Gastroenterology O.O.Bogomolets NMU, Kyiv
  - CI of Kyiv RC Regional Clinical Hospital #2, Kyiv
  - Kyiv CCH #8 Dept of Gastroenterology P.L. Shupyk NMA of PGE, Kyiv
  - Kyiv CCH #18 Dept of Proctology O. O. Bogomolets NMU, Kyiv
  - Lviv Regional Clinical Hospital, Lviv
  - Communal City Clinical Hospital of Ambulance, Dept of Therapy #1 D.Halytskyi Lviv NMU, Lviv
  - CI Sumy City Clinical Hospital #1 Dept of Therapy Sumy SU, Sumy
  - Sumy Regional Clinical Hospital, Sumy
  - CI of TRC Ternopil University Hospital, Ternopil
  - A. Novak Transcarpathian Regional Clinical Hospital, Uzhhorod
  - MCIC MC LLC Health Clinic, Vinnytsia
  - Vinnytsia Regional Clinical Hospital for Invalids of the Great Patriotic War, Vinnytsia
  - M.I. Pyrogov VRCH Dept of Gastroenterology M.I. Pyrogov VNMU, Vinnytsia
  - Vinnytsia M.I. Pyrohov Regional Clinical Hospital, Vinnytsia
  - Vinnytsia M.I. Pyrohov National Medical University, Vinnytsia
  - City Clinical Hospital of Emergency and Urgent Care of Zaporizhzhya, Zaporizhia
  - Zaporizhia City Multispecialty Clinical Hospital #9, Department of Neurology, Zaporizhia
  - CI City Hospital #1, Zaporizhia
  - CI Zapor City Multifunctional CH#9 City Center of Gastroenterology SI Zapor MA of PGE of MOHU, Zaporizhzhia
  - Zaporizhia Regional Clinical Hospital, Zaporizhzhia
  - Central District Hospital under Zhytomyr District Council, Zhytomyr
- United Kingdom (6):
  - University Hospital Coventry, Coventry
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Gloucestershire Royal Hospital, Gloucester
  - Whipps Cross University Hospital, London
  - St Thomas' Hospital, London
  - Royal Shrewsbury Hospital, Shrewsbury

REFERENCES:
- [Derived] Yarur A, Irving P, Siegmund B, Dubinsky MC, Ananthakrishnan AN, Regueiro M, Ungaro RC, Ritter T, Nakase H, Liu Z, Mehra D, Osterman MT, Jain A, Rubin DT, Hibi T. Long-Term Ozanimod Therapy in Patients With Moderately Active Ulcerative Colitis After Failure of 5-Aminosalicylic Acid. Inflamm Bowel Dis. 2026 Jan 1;32(1):77-86. doi: 10.1093/ibd/izaf195. PMID 41003640
- [Derived] Sands BE, Rubin DT, Loftus EV Jr, Wolf DC, Panaccione R, Colombel JF, Dignass A, Regueiro M, Vermeire S, Afzali A, Lawlor G, Ahmad HA, Wu H, Osterman MT, Jain A, D'Haens G. Impact of Prior Biologic Exposure on Ozanimod Efficacy and Safety in the Phase 3 True North Clinical Trial. Am J Gastroenterol. 2025 Oct 1;120(10):2339-2349. doi: 10.14309/ajg.0000000000003310. Epub 2025 Jan 8. PMID 39773524
- [Derived] Regueiro M, Siegmund B, Horst S, Moslin R, Charles L, Petersen A, Tatosian D, Wu H, Lawlor G, Fischer M, D'Haens G, Colombel JF. Concomitant Administration of Ozanimod and Serotonergic Antidepressants in Patients With Ulcerative Colitis or Relapsing Multiple Sclerosis. Inflamm Bowel Dis. 2025 Apr 10;31(4):1010-1017. doi: 10.1093/ibd/izae136. PMID 39018016
- [Derived] Sands BE, D'Haens G, Panaccione R, Regueiro M, Ghosh S, Hudesman D, Ahmad HA, Mehra D, Wu H, Jain A, Petersen A, Osterman MT, Afzali A, Danese S. Ozanimod in Patients With Moderate to Severe Ulcerative Colitis Naive to Advanced Therapies. Clin Gastroenterol Hepatol. 2024 Oct;22(10):2084-2095.e4. doi: 10.1016/j.cgh.2024.03.042. Epub 2024 May 8. PMID 38723981
- [Derived] Armuzzi A, Cross RK, Lichtenstein GR, Hou J, Deepak P, Regueiro M, Wolf DC, Akukwe L, Ahmad HA, Jain A, Kozinn M, Wu H, Petersen A, Charles L, Long M. Cardiovascular Safety of Ozanimod in Patients With Ulcerative Colitis: True North and Open-Label Extension Analyses. Clin Gastroenterol Hepatol. 2024 May;22(5):1067-1076.e3. doi: 10.1016/j.cgh.2023.11.018. Epub 2023 Nov 30. PMID 38040274
- [Derived] Sandborn WJ, Feagan BG, D'Haens G, Wolf DC, Jovanovic I, Hanauer SB, Ghosh S, Petersen A, Hua SY, Lee JH, Charles L, Chitkara D, Usiskin K, Colombel JF, Laine L, Danese S; True North Study Group. Ozanimod as Induction and Maintenance Therapy for Ulcerative Colitis. N Engl J Med. 2021 Sep 30;385(14):1280-1291. doi: 10.1056/NEJMoa2033617. PMID 34587385

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1012 Participants randomized and treated
Groups:
- RPC1063 Cohort 1 (Induction Period): * Blinded
  * On Days 1 to 4, RPC1063/ozanimod HCl 0.25 mg (equivalent to ozanimod 0.23 mg) or matching placebo once daily (one 0.25 mg capsule)
  * On Days 5 to 7, RPC1063/ozanimod HCl 0.5 mg (equivalent to ozanimod 0.46 mg) or matching placebo once daily (two 0.25 mg capsules)
  * On Day 8, patients will receive the final dose RPC1063/ozanimod HCl 1 mg (equivalent to ozanimod 0.92 mg) or matching placebo once daily for 9 weeks (one 1 mg capsule)
- Placebo Cohort 1 (Induction Period): -Blinded Placebo Participants started in induction period and some continued to receive placebo in the Maintenance Period in a double blind manner.
- RPC1063 Cohort 2 (Induction Period): * Open Label
  * On Days 1 to 4, RPC1063/ozanimod HCl 0.25 mg (equivalent to ozanimod 0.23 mg) or matching placebo once daily (one 0.25 mg capsule)
  * On Days 5 to 7, RPC1063/ozanimod HCl 0.5 mg (equivalent to ozanimod 0.46 mg) or matching placebo once daily (two 0.25 mg capsules)
  * On Day 8, patients will receive the final dose RPC1063/ozanimod HCl 1 mg (equivalent to ozanimod 0.92 mg) or matching placebo once daily for 9 weeks (one 1 mg capsule)
- RPC1063 (Maintenance Period): - Blinded RPC1063/ozanimod HCl 1 mg (equivalent to ozanimod 0.92 mg) once daily for 42 weeks (one 1 mg capsule)
- Placebo (Maintenance Period): - Blinded Placebo
Period: Overall Study
Arm/Group | RPC1063 Cohort 1 (Induction Period) | Placebo Cohort 1 (Induction Period) | RPC1063 Cohort 2 (Induction Period) | RPC1063 (Maintenance Period) | Placebo (Maintenance Period)
Started | 429 | 216 | 367 | 0 | 0
Transition to Maintenance Period (Completed Induction Week 10, continuing into MP) | 233 | 69 | 224 | 0 | 0
Treated in Maintenance Period (Subjects who entered Maintenance Period from Induction period) | 0 | 69 | 0 | 230 (Randomized from cohort 1 and 2 RCP1063 treatment) | 227 (Randomized from cohort 1 and 2 RCP1063 treatment)
Completed | 401 | 192 | 324 | 0 | 0
Not Completed | 28 | 24 | 43 | 0 | 0
Not completed — non compliance with protocol | 2 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 11 | 6 | 12 | 0 | 0
Not completed — Lack of Efficacy | 4 | 10 | 9 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 8 | 20 | 0 | 0
Not completed — Other Reason | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- RPC1063 Cohort 1(Induction Period): * Blinded
  * On Days 1 to 4, RPC1063/ozanimod HCl 0.25 mg (equivalent to ozanimod 0.23 mg) once daily (one 0.25 mg capsule)
  * On Days 5 to 7, RPC1063/ozanimod HCl 0.5 mg (equivalent to ozanimod 0.46 mg) once daily (two 0.25 mg capsules)
  * On Day 8, patients will receive the final dose RPC1063/ozanimod HCl 1 mg (equivalent to ozanimod 0.92 mg) once daily for 9 weeks (one 1 mg capsule)
- Total: Total of all reporting groups
Arm/Group | RPC1063 Cohort 1(Induction Period) | Placebo Cohort 1 (Induction Period) | RPC1063 Cohort 2 (Induction Period) | RPC1063 (Maintenance Period) | Placebo (Maintenance Period) | Total
Number analyzed (Participants) | 429 | 216 | 367 | 230 | 227 | 1469
Age, Categorical [Count of Participants; unit: Participants] — Population: Two different periods
  Participants
    Induction Period: number analyzed (Participants) | 429 | 216 | 367 | 0 | 0 | 1012
    Induction Period: <=18 years | 0 | 0 | 0 |  |  | 0
    Induction Period: Between 18 and 65 years | 410 | 202 | 346 |  |  | 958
    Induction Period: >=65 years | 19 | 14 | 21 |  |  | 54
    Maintenance Period: number analyzed (Participants) | 0 | 0 | 0 | 230 | 227 | 457
    Maintenance Period: <=18 years |  |  |  | 0 | 0 | 0
    Maintenance Period: Between 18 and 65 years |  |  |  | 217 | 215 | 432
    Maintenance Period: >=65 years |  |  |  | 13 | 12 | 25
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two different periods
  Participants
    Induction Period: number analyzed (Participants) | 429 | 216 | 367 | 0 | 0 | 1012
    Induction Period: Female | 184 | 73 | 153 |  |  | 410
    Induction Period: Male | 245 | 143 | 214 |  |  | 602
    Maintenance Period: number analyzed (Participants) | 0 | 0 | 0 | 230 | 227 | 457
    Maintenance Period: Female |  |  |  | 117 | 122 | 239
    Maintenance Period: Male |  |  |  | 113 | 105 | 218
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two different periods
  Participants
    Induction Period: number analyzed (Participants) | 429 | 216 | 367 | 0 | 0 | 1012
    Induction Period: Hispanic or Latino | 26 | 8 | 16 |  |  | 50
    Induction Period: Not Hispanic or Latino | 403 | 208 | 351 |  |  | 962
    Induction Period: Unknown or Not Reported | 0 | 0 | 0 |  |  | 0
    Maintenance Period: number analyzed (Participants) | 0 | 0 | 0 | 230 | 227 | 457
    Maintenance Period: Hispanic or Latino |  |  |  | 9 | 13 | 22
    Maintenance Period: Not Hispanic or Latino |  |  |  | 221 | 214 | 435
    Maintenance Period: Unknown or Not Reported |  |  |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two different periods
  Participants
    Induction Period: number analyzed (Participants) | 429 | 216 | 367 | 0 | 0 | 1012
    Induction Period: American Indian or Alaska Native | 0 | 0 | 0 |  |  | 0
    Induction Period: Asian | 36 | 17 | 12 |  |  | 65
    Induction Period: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  |  | 0
    Induction Period: Black or African American | 14 | 4 | 10 |  |  | 28
    Induction Period: White | 370 | 192 | 336 |  |  | 898
    Induction Period: More than one race | 0 | 0 | 0 |  |  | 0
    Induction Period: Unknown or Not Reported | 9 | 3 | 9 |  |  | 21
    Maintenance Period: number analyzed (Participants) | 0 | 0 | 0 | 230 | 227 | 457
    Maintenance Period: American Indian or Alaska Native |  |  |  | 0 | 0 | 0
    Maintenance Period: Asian |  |  |  | 13 | 12 | 25
    Maintenance Period: Native Hawaiian or Other Pacific Islander |  |  |  | 0 | 0 | 0
    Maintenance Period: Black or African American |  |  |  | 9 | 9 | 18
    Maintenance Period: White |  |  |  | 205 | 202 | 407
    Maintenance Period: More than one race |  |  |  | 0 | 0 | 0
    Maintenance Period: Unknown or Not Reported |  |  |  | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Clinical Remission at 10 Weeks
Description: Percentage of participants that are in Clinical remission at 10 weeks
Time Frame: At 10 Weeks
Population: ITT Population
Measure: Number; unit: Percentage
Arm/Group | RPC1063 Cohort 1(Induction Period) | Placebo Cohort 1 (Induction Period) | RPC1063 Cohort 2 (Induction Period) | RPC1063 (Maintenance Period) | Placebo (Maintenance Period)
Number analyzed (Participants) | 429 | 216 | 367 | 0 | 0
Percentage | 18.4 | 6.0 | 21.0 |  |
Statistical Analysis 1: Comparison: RPC1063 Cohort 1(Induction Period) vs Placebo Cohort 1 (Induction Period); Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.586, 95% CI 2-sided [1.938 to 6.636]

2. Primary Outcome: Percentage of Participants in Clinical Remission at 52 Weeks
Description: Percentage of participants that are in Clinical remission at 52 weeks
Time Frame: At 52 Weeks
Population: ITT Population
Measure: Number; unit: Percentage
Arm/Group | RPC1063 Cohort 1(Induction Period) | Placebo Cohort 1 (Induction Period) | RPC1063 Cohort 2 (Induction Period) | RPC1063 (Maintenance Period) | Placebo (Maintenance Period)
Number analyzed (Participants) | 0 | 69 | 0 | 230 | 227
Percentage |  | 24.6 |  | 37.0 | 18.5
Statistical Analysis 1: Comparison: RPC1063 (Maintenance Period) vs Placebo (Maintenance Period); Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.755, 95% CI 2-sided [1.767 to 4.294]

3. Secondary Outcome: Percentage of Participants With Clinical Response at 10 Weeks
Description: Percentage of participants that are in Clinical response at 10 weeks
Time Frame: At 10 Weeks
Population: ITT Population
Measure: Number; unit: Percentage
Arm/Group | RPC1063 Cohort 1(Induction Period) | Placebo Cohort 1 (Induction Period) | RPC1063 Cohort 2 (Induction Period) | RPC1063 (Maintenance Period) | Placebo (Maintenance Period)
Number analyzed (Participants) | 429 | 216 | 367 | 0 | 0
Percentage | 47.8 | 25.9 | 52.6 |  |

4. Secondary Outcome: Percentage of Participants With Endoscopic Improvement at 10 Weeks
Description: Percentage of participants with endoscopic improvement at 10 weeks
Time Frame: At 10 Weeks
Population: ITT Population
Measure: Number; unit: Percentage
Arm/Group | RPC1063 Cohort 1(Induction Period) | Placebo Cohort 1 (Induction Period) | RPC1063 Cohort 2 (Induction Period) | RPC1063 (Maintenance Period) | Placebo (Maintenance Period)
Number analyzed (Participants) | 429 | 216 | 367 | 0 | 0
Percentage | 27.3 | 11.6 | 27.2 |  |

5. Secondary Outcome: Percentage of Participants With Mucosal Healing at 10 Weeks
Description: Percentage of participants with mucosal healing at 10 weeks
Time Frame: At 10 Weeks
Population: ITT Population
Measure: Number; unit: Percentage
Arm/Group | RPC1063 Cohort 1(Induction Period) | Placebo Cohort 1 (Induction Period) | RPC1063 Cohort 2 (Induction Period) | RPC1063 (Maintenance Period) | Placebo (Maintenance Period)
Number analyzed (Participants) | 429 | 216 | 367 | 0 | 0
Percentage | 12.6 | 3.7 | 11.4 |  |

6. Secondary Outcome: Percentage of Participants in Clinical Response at 52 Weeks
Description: Percentage of participants that are in Clinical response at 52 weeks
Time Frame: At 52 Weeks
Population: ITT Population
Measure: Number; unit: Percentage
Arm/Group | RPC1063 Cohort 1(Induction Period) | Placebo Cohort 1 (Induction Period) | RPC1063 Cohort 2 (Induction Period) | RPC1063 (Maintenance Period) | Placebo (Maintenance Period)
Number analyzed (Participants) | 0 | 69 | 0 | 230 | 227
Percentage |  | 39.1 |  | 60.0 | 41.0

7. Secondary Outcome: Percentage of Participants With Endoscopic Improvement at 52 Weeks
Description: Percentage of participants with endoscopic improvement at 52 weeks
Time Frame: At 52 Weeks
Population: ITT Population
Measure: Number; unit: Percentage
Arm/Group | RPC1063 Cohort 1(Induction Period) | Placebo Cohort 1 (Induction Period) | RPC1063 Cohort 2 (Induction Period) | RPC1063 (Maintenance Period) | Placebo (Maintenance Period)
Number analyzed (Participants) | 0 | 69 | 0 | 230 | 227
Percentage |  | 29.0 |  | 45.7 | 26.4

8. Secondary Outcome: Percentage of Participants in Clinical Remission at Week 52 Who Were in Remission at Week 10
Description: Percentage of participants in clinical remission at week 52 who were in clinical remission at week 10
Time Frame: At 52 Weeks
Population: ITT Population who were in remission at week 10
Measure: Number; unit: Percentage
Arm/Group | RPC1063 Cohort 1(Induction Period) | Placebo Cohort 1 (Induction Period) | RPC1063 Cohort 2 (Induction Period) | RPC1063 (Maintenance Period) | Placebo (Maintenance Period)
Number analyzed (Participants) | 0 | 12 | 0 | 79 | 75
Percentage |  | 41.7 |  | 51.9 | 29.3

9. Secondary Outcome: Percentage of Participants With Corticosteroid Free Remission at 52 Weeks
Description: Percentage of participants with corticosteroid free remission at 52 weeks
Time Frame: At 52 Weeks
Population: ITT Population
Measure: Number; unit: Percentage
Arm/Group | RPC1063 Cohort 1(Induction Period) | Placebo Cohort 1 (Induction Period) | RPC1063 Cohort 2 (Induction Period) | RPC1063 (Maintenance Period) | Placebo (Maintenance Period)
Number analyzed (Participants) | 0 | 69 | 0 | 230 | 227
Percentage |  | 24.6 |  | 31.7 | 16.7

10. Secondary Outcome: Percentage of Participants With Mucosal Healing at 52 Weeks
Description: Percentage of participants with Mucosal Healing at 52 weeks
Time Frame: At 52 Weeks
Population: ITT Population
Measure: Number; unit: Percentage
Arm/Group | RPC1063 Cohort 1(Induction Period) | Placebo Cohort 1 (Induction Period) | RPC1063 Cohort 2 (Induction Period) | RPC1063 (Maintenance Period) | Placebo (Maintenance Period)
Number analyzed (Participants) | 0 | 69 | 0 | 230 | 227
Percentage |  | 10.1 |  | 29.6 | 14.1

11. Secondary Outcome: Percentage of Participants With Durable Clinical Remission at 52 Weeks
Description: Percentage of participants with durable clinical remission at 52 weeks
Time Frame: At 52 Weeks
Population: ITT Population
Measure: Number; unit: Percentage
Arm/Group | RPC1063 Cohort 1(Induction Period) | Placebo Cohort 1 (Induction Period) | RPC1063 Cohort 2 (Induction Period) | RPC1063 (Maintenance Period) | Placebo (Maintenance Period)
Number analyzed (Participants) | 0 | 69 | 0 | 230 | 227
Percentage |  | 7.2 |  | 17.8 | 9.7

ADVERSE EVENTS:
Time Frame: Approximately up to 52 Weeks
Description: Participant overlap due to re randomization occuring before maintenance phase
Groups:
- Cohort 1 (Induction Period): RPC1063 1mg: Cohort 1 (Induction Period): RPC1063 1mg
- Cohort 1: Placebo: Cohort 1: Placebo
- Cohort 2 (Induction Period): RPC1063 1mg: Cohort 2 (Induction Period): RPC1063 1mg
- Intervention (Maintenance Period): RPC1063 1mg: Intervention (Maintenance Period): RPC1063 1mg
- Placebo (Maintenance Period): Placebo: Placebo (Maintenance Period): Placebo
Arm/Group | Cohort 1 (Induction Period): RPC1063 1mg | Cohort 1: Placebo | Cohort 2 (Induction Period): RPC1063 1mg | Intervention (Maintenance Period): RPC1063 1mg | Placebo (Maintenance Period): Placebo
All-Cause Mortality (participants affected / at risk) | 0/429 | 0/216 | 1/367 | 0/230 | 0/227
Serious Adverse Events (participants affected / at risk) | 17/429 | 11/216 | 23/367 | 12/230 | 18/227
Other Adverse Events (participants affected / at risk) | 15/429 | 13/216 | 15/367 | 2/230 | 4/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Induction Period): RPC1063 1mg (N=429) | Cohort 1: Placebo (N=216) | Cohort 2 (Induction Period): RPC1063 1mg (N=367) | Intervention (Maintenance Period): RPC1063 1mg (N=230) | Placebo (Maintenance Period): Placebo (N=227)
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 6 | 5 | 9 | 1 | 9
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Proctitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 2 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Complicated appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Large intestine infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Measles (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Yersinia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus test positive (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Induction Period): RPC1063 1mg (N=429) | Cohort 1: Placebo (N=216) | Cohort 2 (Induction Period): RPC1063 1mg (N=367) | Intervention (Maintenance Period): RPC1063 1mg (N=230) | Placebo (Maintenance Period): Placebo (N=227)
Anaemia (Blood and lymphatic system disorders) | 15 | 13 | 15 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT02435992/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT02435992/SAP_001.pdf